CLINICAL TRIAL: NCT05616936
Title: Evaluation of Different Orthodontic Tooth Movements Assisted With Injectable Platelet Rich Fibrin: A Prospective Clinical Study
Brief Title: Evaluation of Different Orthodontic Tooth Movements Assisted With Injectable Platelet Rich Fibrin
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, farouk ahmed hussein, Principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 837/140
Record Dates: First submitted 2022-11-09; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Effect of Platelet Rich Fibrin With Different Tooth Movements

STUDY DESIGN:
Intervention Model Description: Factorial Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group I (Experimental): Intervention side: application of i-PRF with distalization of maxillary first molar that will be performed on intervention sides according to a standardized protocol.
  Interventions: Biological: injectable platelet rich fibrin
- Group II (No Intervention): Control side: distalization of maxillary first molar that will be performed without any intervention
- Group A (Experimental): levelling and alignment assisted with Injectable Platelet-rich fibrin (i-PRF) according to a standardized protocol.
  Interventions: Biological: injectable platelet rich fibrin
- Group B (No Intervention): leveling and alignment will be commenced without Injection of Injectable platelet-rich fibrin (i-PRF)
- Group a (Experimental): Will includes 9 patients who will receive intrusive arch after leveling and alignment assisted Injectable Platelet-rich fibrin (i-PRF) according to a standardized protocol.
  Interventions: Biological: injectable platelet rich fibrin
- Group b (No Intervention): Will includes 9 patients who will receive intrusive utility arches after leveling and alignment without Injection of Injectable platelet-rich fibrin (i-PRF)

INTERVENTIONS:
Biological: injectable platelet rich fibrin — injectable platelet rich fibrin
  Arms: Group A; Group I; Group a

SUMMARY:
The present prospective clinical study will be undertaken for assessment of the effect of application of i-PRF on the rate of levelling and alignment, molar distalization& intrusion of anterior teeth in deep bite cases

DETAILED DESCRIPTION:
Assessment of the effect of application of i-PRF on the rate of levelling and alignment, molar distalization& intrusion of anterior teeth in deep bite cases

ELIGIBILITY:
Inclusion Criteria:An age range from 15-22 years. Severe crowding or protrusion requiring 1st premolars extractions followed by symmetrical canine retraction.

All permanent teeth present, 3rd molars are excluded. Good oral and general health. No systemic disease/medication that could interfere with orthodontic tooth movement. No previous orthodontic treatment.

-

Exclusion Criteria:Patient diagnosed to have an indication for non-extraction approach.

Poor oral hygiene or periodontally compromised patient. Patient with craniofacial anomalies or previous history of trauma, bruxism or parafunctions.

-

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
effect of injectable platelet rich fibrin on different tooth movements | post interventional at 4 months
  rate of tooth movement

CONTACTS AND LOCATIONS:
Locations (1):
- AlAzhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Effect of injectable platelet-rich fibrin (i-PRF) in accelerating orthodontic tooth movement : A randomized split-mouth-controlled trial. J Orofac Orthop. 2021 Jul;82(4):268-277. doi: 10.1007/s00056-020-00275-x. Epub 2021 Jan 22. PMID 33481053
- [Background] Erdur EA, Karakasli K, Oncu E, Ozturk B, Hakki S. Effect of injectable platelet-rich fibrin (i-PRF) on the rate of tooth movement. Angle Orthod. 2021 May 1;91(3):285-292. doi: 10.2319/060320-508.1. PMID 33459765